CLINICAL TRIAL: NCT04362202
Title: A Water-based Sequential Preparatory Approach Versus Conventional Aquatic Training in Stroke Patients: a Randomized Controlled Trial With a One-month Follow-up
Brief Title: A Water-based Sequential Preparatory Approach and Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Marco Tramontano, Head of Rehabilitation Services, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FSLCE/PROG.728
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): 8 individual experimental rehabilitation sessions as outpatients (2 days/week, 4 weeks), in a rehabilitation pool at Fondazione Santa Lucia Neurorehabilitation hospital. Each session lasted 45minutes. The water temperature was between 30°C and 32°C.
  Interventions: Other: Water-based Sequential Preparatory Approach
- control (Active Comparator): 8 individual of standard aquatic rehabilitation sessions as outpatients (2 days/week, 4 weeks), in a rehabilitation pool at Fondazione Santa Lucia Neurorehabilitation hospital. Each session lasted 45minutes. The water temperature was between 30°C and 32°C.
  Interventions: Other: Water-based Sequential Preparatory Approach

INTERVENTIONS:
Other: Water-based Sequential Preparatory Approach — The experimental training consists of a sequential and a preparatory approach aimed at enhancing dynamic postural stability. The exercises followed a specific sequence starting from a kneeling position, proceeding to a sitting position and ending with a supine position. Step exercises preparatory for gait were performed using a step and two floating aids. Gait exercises were performed first with the upper limbs placed on two floating aids and then during a dual motor task (i.e., catching a ball thrown by the therapist).
  The control aquatic therapy consists of water-based exercises, in line with suggestions of the Hydrotherapy Association of Chartered Physiotherapists Guidance on Good Practice in Hydrotherapy.
  These consisted of warm-up exercises, stretching exercises for the lower limbs, recruitment exercises and walking exercises during each phase of gait (single stance, swing and double stance).

SUMMARY:
Many studies hypothesize that people who have suffered stroke could benefit from water-based exercises to improve their strength and ability to perform the activities of daily living.

A Cochrane Review systematically synthesized and compared the effects of aquatic and land-based therapies on the activities of daily living (ADL) of patients following stroke and found that water-based exercises improved strength and ADL. A recent review indicates that RCTs comparing aquatic methods in both environments are lacking. The same movements in water and on dry land that target postural stability and gait require different competences. For example, the postural instability that occurs while squatting in water was enacted on land by sitting on a therapy ball. Furthermore, land-based conventional rehabilitation is generally task oriented, customized and challenging and follows a specific preparatory sequence of exercises according to patients' disabilities. Therefore, the investigators believe that a sequential preparatory approach (SPA), based on increasing difficulty and following a specific sequence of preparatory exercises (from the simplest to the most complex), should also be used in an aquatic environment.

ELIGIBILITY:
Inclusion Criteria:

* Stroke with unilateral hemiplegia within the previous six months;
* Ability to walk without any device or need of continuous physical assistance to support body weight or maintain balance (Functional Ambulation Classification ≥ 3);
* Acclimatization to water.

Exclusion criteria:

* Cognitive deficits affecting the ability to understand task instructions (Mini-Mental State Examination > 24);
* Severe unilateral spatial neglect (diagnosed with a test battery that included the Letter Cancellation test, Barrage test, Sentence Reading test and the Wundt-Jastrow Area Illusion Test);
* Severe aphasia (diagnosed by means of neuropsychological assessment);
* Presence of other neurological diseases;
* Presence of cutaneous and mycosis infections;
* Presence of open wounds, eczema, skin ulcers, decubitus lesions, severe burns;
* Presence of PEG (Percutaneous endoscopic gastrostomy);
* Presence of tracheostomy;
* Urinary incontinence;
* Presence of otitis
* Presence of orthopedic or cardiac comorbidities that would limit participation in the experimental and conventional training (all of which were clinically evaluated).

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Berg Balance Scale at 2 months | at 2 months
  Change of Berg Balance Scale (BBS) from baseline at 2 months. BBS values ranging from 0 to 56, where 0 means the lowest level of function and 56 the highest

SECONDARY OUTCOMES:
Stroke Specific Quality Of Life Scale (SS-QOL) | baseline, after 4 weeks of training, and 4 weeks after the end of training
  Change of Stroke Specific Quality Of Life Scale (SS-QOL) from baseline at 4 weeks of training and at 4 weeks after the end of the training. SS-QOL values ranging from 0 to 245, where 0 means the worse outcome and 245 the best one.
Modified Barthel Index (MBI) | baseline, after 4 weeks of training, and 4 weeks after the end of training
  Change of Modified Barthel Index (MBI) from baseline at 4 weeks of training and at 4 weeks after the end of the training. MBI values ranging from 0 to 105, where 0 means the worse outcome and 105 the best one.
Tinetti Balance and Gait Scale (TBG) | baseline, after 4 weeks of training, and 4 weeks after the end of training
  Change of Tinetti Balance and Gait Scale (TBG) from baseline at 4 weeks of training and at 4 weeks after the end of the training. TBG values ranging from 0 to 28, where 0 means the worse outcome and 28 the best one.
Modified Ashworth Scale (MAS) | baseline, after 4 weeks of training, and 4 weeks after the end of training
  Change of Modified Ashworth Scale (MAS) from baseline at 4 weeks of the training and at 4 weeks after the end of the training. MAS values ranging from 0 to 5, where 0 means the best outcome and 5 the worse one.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Tramontano, Principal Investigator — Santa Lucia Foundation I.R.C.C.S.
Locations (1):
- Santa Lucia Foundation I.R.C.C.S., Roma, Rm, Italy